CLINICAL TRIAL: NCT04740736
Title: Cardiovascular Analysis of Post-exertional Malaise
Brief Title: Cardiovascular Analysis of PEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Benjamin Natelson, Professor, Neurology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 19-1952; R01NS117638 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline Infusion (Experimental)
  Interventions: Procedure: Saline Infusion
- Sham Infusion (Sham Comparator)
  Interventions: Procedure: Saline Infusion

INTERVENTIONS:
Procedure: Saline Infusion — Patient with hypovolemia on day 1 will be randomized to a saline or sham infusion prior to the Day 2 exercise test.

SUMMARY:
The purpose of this study is to examine cardiopulmonary function in Chronic Fatigue Syndrome (CFS) patients and determine how it relates to the common symptom of Post-exertional malaise (PEM). Subjects will complete a maximal exercise test on 2 subsequent days. Total blood volume will be measured prior to each exercise test, and patient with hypovolemia on day 1, will be randomized to either a saline or sham infusion prior to the 2nd exercise test. A total of 80 CFS patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25 to 60
* Meet the 2015 IOM case definition for ME/CFS

Exclusion Criteria:

* Patients with a medical cause for their fatigue
* Patients taking medications that would dampen cardiac response to exercise
* Patients with psychotic illness, bipolar disorder, or current major depressive disorder
* Patients with a history of anorexia or bulimia within 5 years of intake
* Patients with a history of alcohol or drug abuse within 2 years of intake

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
CPET testing | 2 days
  To assess VO2VT and peak VO2
Total Blood Volume | 2 days
  To measure Total Blood Volume (TBV) before each exercise test
Hypovolemia | 1 day
  Patients with reduced Total Blood Volume on day #1 CPET will be randomized in a 1:1 fashion to either a one hour infusion of a liter of isotonic saline prior to day #2 CPET or a sham infusion

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Natelson, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/36/NCT04740736/ICF_000.pdf